CLINICAL TRIAL: NCT04867798
Title: Transgender Men and HIV in Uganda: PrEP Uptake and Persistence
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REC REF 1208-2020
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: HIV; Sexually Transmitted Infections; PrEP; Transgender Men
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lamivudine-Tenofovir 300 Mg-300 Mg Oral Tablet — PrEP eligible participants will be asked to follow up monthly for 12 months. PrEP will be prescribed for once-daily use and discontinued if HIV tests are positive. At quarterly visits, participants will receive Integrated Next Steps Counseling (iNSC) for PrEP adherence with point-of-care drug level feedback. Participants will receive iNSC Support Level 1 to address PrEP adherence and sexual health needs. Those with urine tenofovir levels <1500 ng/mL will receive iNSC Support Level 2, in which participant responses to two 7-item questionnaires on PrEP adherence and sexual health will guide problem solving on improved dosing. Medication refills will consist of 3-month supplies.

SUMMARY:
Transgender men (trans men; assigned female sex at birth but identify as male) are generally thought to be at low risk of HIV acquisition, perhaps because of the assumption that they have sex with cis-gender women. Emerging data from resource-rich settings show that trans men often face many of the same high risks as transgender women (trans women; assigned male sex at birth but identify as female). Trans men report similar rates to trans women of engagement in sex work and engage in unprotected receptive vaginal and/or anal sex with cis-gender men. Additionally, they report high sexual risk-taking behaviors including inconsistent condom use which puts them at risk of HIV and other sexually transmitted infections (STIs). Little is known about HIV risk in trans men globally, and no published data are available from sub-Saharan Africa. We will recruit a cohort of 50 trans men through respondent driven sampling. We will use mixed methods to gain a deeper understanding of the sexual health experiences and risk behaviors of trans men in Uganda. Guided by the Social Ecological Model, we will conduct in-depth interviews with up to 20 trans men to understand individual, interpersonal, community and social contextual factors that influence sexual risk behaviors and HIV/STI risk (Aim 1). In Aim 2, we will characterize HIV and STI prevalence and risk among trans men by conducting a behavioral HIV risk assessment including sexual practices, alcohol and drug use, partner violence, gender dysphoria, male hormone use and willingness to take PrEP. In Aim 3, we will evaluate PrEP uptake and persistence among HIV-negative trans men with HIV risk. Participants will be offered PrEP and followed monthly for 12 months. At quarterly visits, participants will receive integrated next steps adherence counseling and drug level feedback using a point-of-care urine tenofovir lateral-flow immunoassay. Free testing and treatment of common curable STIs (Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis) will be provided. Primary outcomes are: 1) PrEP persistence at 6 and 12 months as measured by tenofovir levels in dried blood spots collected quarterly, and 2) STI incidence. Assessment of PrEP use by trans men will help increase the utilization of HIV services, including HIV and STI testing and PrEP, with a goal of decreasing HIV acquisition.

DETAILED DESCRIPTION:
Transgender men (trans men; assigned female sex at birth but identify as male) are generally thought to be at low risk of HIV acquisition, perhaps because of the assumption that they have sex with cis-gender women. Emerging data from resource-rich settings show that trans men often face many of the same high risks as transgender women (trans women; assigned male sex at birth but identify as female). Trans men report similar rates to trans women of engagement in sex work and engage in unprotected receptive vaginal and/or anal sex with cis-gender men. Additionally, they report high sexual risk-taking behaviors including inconsistent condom use which puts them at risk of HIV and other sexually transmitted infections (STIs). Little is known about HIV risk in trans men globally, and no published data are available from sub-Saharan Africa. In partnership with the trans community, we are testing the effectiveness of peer-delivered HIV self-testing, STI self-sampling and pre-exposure prophylaxis (PrEP) (Peer Study), same-day PrEP initiation and sexual health for trans women in Uganda (Tandika PrEP Study) and conducting a pilot evaluation of HIV and STI risk in trans men (HASTE study). This study is designed to leverage the community linkages, collaborative partnerships with transgender organizations, peer networks, scientific expertise and research infrastructure of these ongoing studies with trans women and men and proposes a concurrent mixed methods study (1) to explore HIV and STI risk characteristics, and PrEP adherence among trans men. Thus, the work extends our unique research experience in the transgender population in Uganda and this study will be the first, to our knowledge, to characterize HIV and STI risk and PrEP adherence among trans men in sub-Saharan Africa.

Approach: In Aim 1, we will characterize HIV and STI prevalence and risk in a new cohort of trans men. In Aim 2, we will evaluate PrEP uptake and persistence among HIV-negative trans men followed for 12 months. In Aim 3, we will explore the sexual health experiences and risk behaviours of trans men.

Aim 1: Characterize HIV and STI prevalence and risk among trans men. We will recruit a novel cohort of up to 50 trans men through the respondent driven sampling (RDS) approaches used in the above-noted studies. We will conduct a behavioral HIV risk assessment including questions about gender identity, HIV and STI testing, and willingness to take PrEP. Interviewer-administered questionnaires will collect data on demographic characteristics, HIV and STI testing behaviors, perception of risk, alcohol and drug use, sexual practices, partner violence, gender dysphoria and male hormone use. Primary outcomes will be: 1) HIV prevalence as measured by the proportion testing HIV positive, 2) STI prevalence as measured by Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis test positivity and 3) sexual risk behaviours as measured by the proportion reporting condom-less sex.

Aim 2: Evaluate PrEP uptake and persistence among HIV-negative trans men. HIV-negative trans men will be offered PrEP and followed monthly for 12 months. At quarterly visits, participants will receive integrated next steps counseling (iNSC) adherence counseling and drug level feedback using a point-of-care (POC) urine tenofovir lateral-flow immunoassay. Free testing and treatment of common curable STIs (Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis) will be provided. Those who screen positive for depression will be actively linked to mental health services. Primary outcomes are: 1) PrEP uptake as measured by pharmacy records and 2) PrEP persistence as measured by intracellular tenofovir diphosphate concentrations in dried blood spots at months 6 and 12.

Aim 3: Explore sexual health experiences and risk behaviours of trans men in Uganda.

We will use qualitative methods to gain a deeper understanding of the sexual health experiences of trans men in the context of their everyday lives and communities. Guided by the Social Ecological Model, we will conduct in-depth interviews with up to 20 trans men to understand individual, interpersonal, community and social contextual factors that influence sexual risk behaviors and HIV/STI risk. We will explore unmet HIV/STI prevention needs, examine perceptions of PrEP and explore barriers and facilitators of retention in HIV care (stigma, discrimination, and concerns about interactions between hormones and PrEP).

ELIGIBILITY:
Inclusion Criteria:

* Report female sex assigned at birth but currently identify as male
* Age ≥18, or if 14-17 years, qualification as a mature or emancipated minor due to having a sexually transmitted infection or cater for own livelihood
* Report condom-less sex in the past 6 months
* Able and willing to provide written informed consent

Exclusion Criteria:

* Currently enrolled in a biomedical HIV prevention study
* Any clinically significant or chronic medical condition that is considered progressive or in the opinion of the investigator would make the participant unsuitable for the study, including severe infections requiring treatment such as tuberculosis, alcohol or drug abuse, or mental illness which preclude provision of informed consent. Those with alcohol or drug abuse who are able to independently provide consent will be not be excluded.
* Not planning to remain in the geographic area for the duration of the study

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identify as transgender men
Study Population: Transgender men (up to 50 participants). Gender identity will be assessed using a two-step approach:
  1. What is your current gender?
  2. What sex were you assigned at birth?
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
PrEP effectiveness as measured by intracellular tenofovir diphosphate levels in dried blood spots | 12 months
  Proportion with tenofovir concentrations ≥700 fmol per punch

SECONDARY OUTCOMES:
Correlates of PrEP adherence as measured by demographic characteristics and sexual behaviors | 12 months
  Association between HIV risk and PrEP adherence

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mujugira, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute Kasangati, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mujugira A, Kasiita V, Bagaya M, Nsubuga R, Nakyanzi A, Nampewo O, Nalumansi A, Kamusiime B, Bambia F, Muwonge TR, Gandhi M, Ware NC, Haberer JE. Oral PrEP Use by Transgender Men in Uganda: A Multi-method Evaluation. AIDS Behav. 2025 Nov 12. doi: 10.1007/s10461-025-04954-x. Online ahead of print. PMID 41222617